CLINICAL TRIAL: NCT07385014
Title: MULTICENTER, DOUBLE-ARM, PATIENT AND ASSESSOR-MASKED, PROSPECTIVE, RANDOMIZED CLINICAL TRIAL TO COMPARE VISUAL PERFORMANCE OF NEGATIVE AND NEUTRAL ASPHERIC MONOFOCAL INTRAOCULAR LENSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Seth M Pantanelli, Professor, Department of Ophthalmology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21065
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cataract; Presbyopia
Keywords: intraocular lens; Presbyopia; Cataract surgery
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Johnson & Johnson Eyhance (Active Comparator): This research is being done to investigate how patients see at far, intermediate, and near distances after cataract surgery
  Interventions: Device: Negative Aspheric Monofocal IOL
- Bausch & Lomb enVista. (Active Comparator): This research is being done to investigate how patients see at far, intermediate, and near distances after cataract surgery
  Interventions: Device: Neutral Aspheric Monofocal IOL

INTERVENTIONS:
Device: Neutral Aspheric Monofocal IOL — IOL implantation following cataract extraction
  Arms: Bausch & Lomb enVista.
Device: Negative Aspheric Monofocal IOL — IOL implantation following cataract extraction
  Arms: Johnson & Johnson Eyhance

SUMMARY:
The purpose of this study is to compare the binocular distance, intermediate, and near visual acuity and patient reported outcomes of the Johnson &Johnson Eyhance and Bausch & Lomb enVista IOLs.

We hypothesize that the Johnson & Johnson's Eyhance and Bausch & Lomb enVista IOLs will have similar distance, intermediate, and near visual acuity.

DETAILED DESCRIPTION:
This research is being done to investigate how patients see at far, intermediate, and near distances after cataract surgery with one of two intraocular lenses: Johnson & Johnson Eyhance or Bausch & Lomb enVista. Note that neither of these lenses are considered investigational devices; both lenses are FDA approved in the United States for implantation during cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 or older at the time of study enrollment.
2. Visually significant cataract in the study eye for which phacoemulsification cataract extraction and posterior chamber IOL implantation is indicated.
3. Projected postoperative CDVA 0.20 logMAR (Snellen 20/32) or better in the study eye, as determined by an Investigator's medical judgement.
4. Calculated spherical power targeted at emmetropia at distance in the study eyes.
5. Calculated IOL power between +5.0 - +34.0 D, inclusive, in both eyes.
6. Measured keratometric astigmatism less than 1.0 D if against-the-rule or 1.5 D if with-the-rule/oblique.
7. If wearing rigid gas permeable (RGP) contact lens in the study eye, willingness to discontinue lens wear for ≥ 21 days prior to preoperative biometry.
8. Availability, willingness, and sufficient cognitive awareness to return for study-required visits and comply with examination procedures.
9. Willingness to sign the IRB-approved informed consent form (ICF) for study participation.

Exclusion Criteria:

1. Mature cataract in the study eye that is likely to prolong surgical procedure and/or lead to intraoperative complications prior to attempted IOL implantation.
2. Any visually significant intraocular media opacity other than cataract in the study eye (as determined by the investigator). Such opacities might include corneal scar or vitreous hemorrhage.
3. Abnormal corneal findings in the study eye (e.g. keratoconus, pellucid marginal degeneration, irregular astigmatism).
4. Any anterior segment pathology in the study eye that could significantly affect outcomes (e.g. chronic uveitis, iritis, aniridia, clinically significant corneal dystrophies, etc.)
5. Any condition in the study eye that could affect IOL stability (e.g. pseudoexfoliation, zonular dialysis, evident zonular weakness or dehiscence, etc.).
6. History of severe dry eye in the study eye that, in the judgement of the investigator, would impair the ability to obtain reliable study measurements.
7. History of serious corneal disease (e.g. herpes simplex, herpes zoster keratitis, etc.) in the study eye.
8. History of any clinically significant retinal pathology or ocular diagnosis in the study eye that could, in the investigator's best judgement, alter or limit final post-operative visual prognosis (e.g. diabetic retinopathy, ischemic disease, macular degeneration, retinal detachment, optic neuropathy, amblyopia, strabismus, aniridia, epiretinal membrane, etc.).
9. History of cystoid macular edema in either eye.
10. History of uveitis in either eye.
11. History of intraocular or corneal surgery in the study eye besides laser peripheral iridotomy (LPI), selective laser trabeculoplasty (SLT), or argon laser trabeculoplasty (ALT).
12. Uncontrolled glaucoma in the study eye (per Investigator judgement).
13. Current ocular infection in the study eye.
14. Presence of uncontrolled systemic disease that could increase operative risk (e.g. diabetes mellitus, mental illness, dementia, clinically significant atopic disease, etc.).
15. Planned concomitant ocular procedure during cataract surgery inclusive of glaucoma surgery e.g. MIGS or limbal relaxing incisions.
16. Unsuitable for study participation for any other reason, as determined by the Investigator's clinical judgement.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 1 month post cataract surgery
  Mean logMAR best-distance corrected visual acuity at intermediate (66 cm) tested in binocular photopic conditions at 1 month (binocular DCIVA).

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All study results